CLINICAL TRIAL: NCT07023666
Title: Early Detection and Management of Cardiac Iron Overload in Sickle Cell Disease Using Multimodal Imaging for Improved Clinical Outcomes
Brief Title: Early Screening and Treatment of Heart Complication in Sickle Cell Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INOVA-2023-159
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Disease
Keywords: Iron Overload; Cardiomyopathies; Arrhythmias
MeSH Terms: conditions — Anemia, Sickle Cell; Iron Overload; Cardiomyopathies; Arrhythmias, Cardiac | interventions — Deferoxamine; Deferasirox; Deferiprone; Echocardiography; Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention for Cardiac Iron Overload in Sickle Cell Patients (Experimental): The study intervention consists of regular cardiac monitoring, iron chelation therapy and guideline-directed medical therapy (GDMT).
  Interventions: Drug: Deferoxamine; Drug: Deferasirox; Drug: Deferiprone; Device: Echocardiography; Device: Electrocardiogram (ECG)

INTERVENTIONS:
Drug: Deferoxamine — Deferoxamine is used to reduce excess iron accumulation after monitoring iron levels. Adjustment to therapy will be based on iron burden assessments throughout the study duration.
  Other Names: Desferal
Drug: Deferasirox — Deferasirox is used for iron chelation therapy based on iron burden assessment throughout the study.
  Other Names: Jadenu, Exjade
Drug: Deferiprone — Deferiprone is used for iron chelation therapy used throughout the study.
  Other Names: Ferriprox
Device: Echocardiography — This device uses ultrasound waves to create images of heart to help evaluate the heart's structure and function. This allows the detection of abnormalities of heart due to iron overload through out the study.
Device: Electrocardiogram (ECG) — The Electrocardiogram (ECG) device records the electrical activity of the heart. It is crucial for identifying arrhythmias and conduction abnormalities, which can be exacerbated by iron accumulation in the heart.

SUMMARY:
This study tests whether early heart screening and treatment for iron overload in subjects with sickle cell disease can prevent heart problems and reduce hospitalizations.

DETAILED DESCRIPTION:
The goal of the study is to detect iron-related heart problems in subjects with sickle cell disease (SCD) through regular cardiac imaging (electrocardiogram, echocardiogram, cardiac MRI) and lab testing every 3 months during the 12 months period. The treatment will be with iron chelation and guideline-directed heart medications.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosis of sickle cell disease (any genotype)
* Serum ferritin levels ≥ 400 ng/mL (up to 80 patients), or less than 400 ng/mL in those who have cardiac symptoms including shortness of breath and lower extremity edema (up to 20 patients)
* Willingness to undergo regular imaging (echocardiograms, ECG, cardiac MRI)
* ECOG performance status of 0-1
* Able to read, understand and provide written informed consent
* Deemed appropriate for participation by the treating physician

Exclusion Criteria:

* Unable to schedule and required follow-up visits
* Medical comorbidities including:
* Known heart failure
* Unstable angina
* Uncontrolled dysrhythmias
* Acute pulmonary embolism
* Active infection or severe comorbid conditions that in the view of the investigator would limit participation
* History of hypersensitivity or contraindication to chelation therapy
* Severe renal or hepatic impairment
* Pregnancy of breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Hospitalization for Sickle Cell Disease Related Complications | Up to 12 months
  Total number of participants hospitalized for SCD related complications including vaso-occlusive crises, acute chest syndrome and infection detect the impact of early intervention of cardiac iron overload in patients with Sickle Cell Disease
Length of Stay for SCD-Related Complications | Up to 12 Months
  The total number of days spent in the hospital per admission for complications related to SCD.

SECONDARY OUTCOMES:
Incidence of Left and/or Right Heart Failure | Up to 12 Months
  Total number of participants who develop left and/or right heart failure is estimated using descriptive statistics with 95% confidence intervals.
Incidence of Atrial or Ventricular Arrhythmia or Conduction Abnormalities | Up to 12 Months
  The number of participants with conditions such as atrial fibrillation, ventricular tachycardia, or conduction system disease. Reported with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Sheinei Alan, MD, Principal Investigator — Inova Fairfax Hospital
Locations (2):
- United States (2):
  - Inova Schar Cancer, Fairfax, Virginia
  - Inova Health Care Service, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzhugh CD, Lauder N, Jonassaint JC, Telen MJ, Zhao X, Wright EC, Gilliam FR, De Castro LM. Cardiopulmonary complications leading to premature deaths in adult patients with sickle cell disease. Am J Hematol. 2010 Jan;85(1):36-40. doi: 10.1002/ajh.21569. PMID 20029950
- [Background] Hamideh D, Alvarez O. Sickle cell disease related mortality in the United States (1999-2009). Pediatr Blood Cancer. 2013 Sep;60(9):1482-6. doi: 10.1002/pbc.24557. Epub 2013 Apr 23. PMID 23637037
- [Background] Lanzkron S, Carroll CP, Haywood C Jr. Mortality rates and age at death from sickle cell disease: U.S., 1979-2005. Public Health Rep. 2013 Mar-Apr;128(2):110-6. doi: 10.1177/003335491312800206. PMID 23450875
- [Background] Whipple NS, Naik RJ, Kang G, Moen J, Govindaswamy SD, Fowler JA, Dowdy J, Penkert R, Joshi VM, Hankins JS. Ventricular global longitudinal strain is altered in children with sickle cell disease. Br J Haematol. 2018 Dec;183(5):796-806. doi: 10.1111/bjh.15607. Epub 2018 Nov 19. PMID 30450553
- [Background] Darbari DS, Sheehan VA, Ballas SK. The vaso-occlusive pain crisis in sickle cell disease: Definition, pathophysiology, and management. Eur J Haematol. 2020 Sep;105(3):237-246. doi: 10.1111/ejh.13430. Epub 2020 May 19. PMID 32301178
- [Background] Modell CB. Haemoglobinopathies. The pathophysiology of beta-thalassaemia major. J Clin Pathol Suppl (R Coll Pathol). 1974;8:12-8. No abstract available. PMID 4536357
- [Background] Taher AT, Saliba AN. Iron overload in thalassemia: different organs at different rates. Hematology Am Soc Hematol Educ Program. 2017 Dec 8;2017(1):265-271. doi: 10.1182/asheducation-2017.1.265. PMID 29222265